CLINICAL TRIAL: NCT04600206
Title: Existential Distress in Patients with Advanced Cancer and Their Caregivers: a Longitudinal Cohort Study
Brief Title: Existential Distress in Patients with Advanced Cancer and Their Caregivers
Status: Completed | Type: Observational
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Sponsor
Other Study IDs: DKH70113404
Record Dates: First submitted 2020-08-29; First posted 2020-10-23 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Neoplasms Malignant; Carcinoma; Palliative Care
Keywords: Advanced cancer; Caregivers; Death anxiety; Demoralization; Existential distress; Longitudinal studies; Mental disorders
MeSH Terms: conditions — Neoplasms; Carcinoma; Necrophobia; Mental Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Patients: Adult patients across all phases of advanced disease (UICC stage IV solid tumor or stage III lung or ovarian tumor) from diagnosis to terminal stages
  Interventions: Other: Self-report questionnaires
- Caregivers: Adult informal caregivers of patients who are diagnosed with stage IV solid tumors or stage III lung or ovarian tumors
  Interventions: Other: Self-report questionnaires

INTERVENTIONS:
Other: Self-report questionnaires — In this longitudinal cohort study, patients and caregivers will not receive an intervention. In addition to the outcomes named in the section "Outcome Measures" patients and caregivers will complete self-report questionnaires for
  Existential distress (Demoralization Scale-II, Death and Dying Distress Scale, Depressive Experiences Questionnaire, Revised Loss Orientation and Life Engagement in Advanced Cancer Scale, Sense of Dignity Item, Patient Dignity Inventory, Marwit-Meuser Caregiver Grief Inventory, Caregiver Guilt Questionnaire)
  Need for and utilization of psychosocial support
  Resources (Sources of Meaning and Meaning in Life Questionnaire, Questionnaire on the Defiant Power of the Human Spirit) and
  Control variables (Memorial Symptom Assessment Scale, PHQ-9 and GAD-7)

SUMMARY:
Despite the potential for alleviation of existential distress through psychosocial interventions, existential concerns and their impact on health care outcomes of patients and caregivers have not yet been systematically studied. The aim of this longitudinal cohort study is to investigate the frequency, longitudinal trajectory and predictive impact of existential distress on patient- and caregiver-relevant end-of-life outcomes. Further, it aims to determine the need for and utilization of psychosocial support in patients and caregivers with regard to existential concerns.

DETAILED DESCRIPTION:
Due to medical progress and an aging population, the number of patients and caregivers who face the profound existential challenges of advanced incurable cancer is constantly growing. Clinically significant existential distress may result from a fear of suffering and perceived lack of control, fear and uncertainty about the end of life, feelings of burdensomeness or insufficiency, grief about missed opportunities, and profound loneliness. Such distress may have a unique and independent contribution to health care outcomes at the end of life. Despite an increasing interest in existential and palliative care interventions that discuss such issues openly, a lack of systematic quantitative data on existential distress and specific support needs hampers clinicians to consequently detect and address existential needs. This longitudinal study aims to 1) systematically investigate the frequency, longitudinal trajectory and predictive impact of existential distress on patient- and caregiver-relevant end-of-life outcomes and 2) determine patients' and caregivers' specific need for and utilization of psychosocial support with respect to existential concerns.

Adult patients diagnosed with advanced cancer and caregivers will be consecutively recruited from outpatient and inpatient treatment facilities of the Univer-sity Cancer Center Hamburg and affiliated clinics. Existential distress, end-of-life outcomes, and mental disorders in 1,000 participants (500 patients, 500 care-givers) will be assessed using self-report questionnaires at five points of assessment over a period of 12 months and diagnostic interviews (at baseline, after six months). To determine the prevalence of existential distress, mental disorders and palliative care outcomes descriptive statistics will be calculated. Descriptive analyses will also be used to examine the need for and utilization of psychosocial support. To investigate the predictive impact of existential distress and patient- and caregiver-relevant end-of-life outcomes multiple linear and logistic regression will be conducted. To analyze longitudinal trajectory of existential distress growth mixture models will be used.

Shaping a clear and systematic knowledge about frequent and persistent existential concerns that are most relevant to the risk for unfavorable end-of-life outcomes, results will significantly contribute to the recognition and manage-ment of existential distress and provide a valuable basis for the development of targeted interventions.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older
* UICC stage IV solid tumor or UICC stage III lung or ovarian tumor
* Informed consent

Exclusion Criteria:

* Severe cognitive
* Severe physical impairment
* Insufficient German to give informed consent and complete self-report questionnaires

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * Patients across all phases of advanced disease from diagnosis to terminal stages who are treated in outpatient and inpatient treatment facilities of the University Cancer Center Hamburg and affiliated clinics
  * Caregivers whose relatives are diagnosed with advanced cancer
Sampling Method: Probability Sample
Enrollment: 800 (Actual)
Dates: Start 2020-10-23 (Actual); Primary Completion 2024-12-08 (Actual); Study Completion 2024-12-08 (Actual)

PRIMARY OUTCOMES:
Aggressiveness of care | 4 weeks prior to death
  Will be assessed for patients according to the criteria by Earle et al., 2003: receipt of chemotherapy in the last two weeks of life, emergency hospital admissions or intensive-care treatment during the last month of life. Will be obtained from medical chart reviews for deceased patients.
Prevalence of affective and anxiety disorders | 6-months follow-up
  Will be assessed for patients and caregivers using the Structured Clinical Interview for Diagnostic and Statistical Manual of Mental Disorders (SCID-5, Beesdo-Baum et al., 2019).
Prevalence of adjustment disorder | 6-months follow-up
  Will be assessed according to International Classification of Diseases (ICD-11) for patients and caregivers using the Adjustment Disorder Module of the CIDI (Composite International Diagnostic Interview, (Perkonigg et al., 2018).
Prevalence of substance use disorders | 6-months follow-up
  Will be assessed for patients and caregivers using the Structured Clinical Interview for Diagnostic and Statistical Manual of Mental Disorders (SCID-5, Beesdo-Baum et al., 2019).
  Will only be assessed for patients and caregivers who were recruited at location no.4 (Specialized Outpatient Clinic for Autoimmune Liver Disease and for Liver and Bile Duct Tumors, University Medical Center Hamburg-Eppendorf).

SECONDARY OUTCOMES:
Desire for hastened death | 6- and 12-months-follow-up
  Will be assessed for patients using the short form of the Schedule of Attitudes Toward Hastened Death (SAHD-A, Kolva et al., 2017). Items are scored with either being true (1) or false (0). The total score is the number of endorsed items, ranging from 0 to 6, with high scores indicating high levels of desire for hastened death.
Suicidal ideation | 6- and 12-months-follow-up
  Will be assessed for patients and caregivers using the Beck Scale for Suicidal Ideation (BSS, Kliem & Brähler, 2015). Items are scored from 0 to 2 (e.g., 0 = I have a moderate to strong wish to live, 1 = I have a weak wish to live, 2 = I have no wish to live). The sum score ranges from 0 to 38 for the total scale, with higher scores indicating stronger suicidal tendencies.
Coping and Demoralization | 6-months follow-up
  Will be assessed for patients and caregivers using the Structured Interview for Psychological Adjustment and Demoralisation (Bobevski & Kissane, 2019). Participants may answer most of the questions with yes or no.
Complicated grief | 3 months post-death
  Will be assessed for caregivers after the patient's death using the Inventory of Complicated Grief (ICG; Lumbeck et al., 2012). Items are scored from 0 (never) to 4 (always). The sum score ranges from 0 to 76, with scores ≥ 25 indicating experiences of complicated grief.
Quality of dying and death | 3 months post-death
  Will be assessed from the caregivers' perspective using a shot version of the Quality of Dying and Death Questionnaire (QODD, Mah et al., 2020). Caregivers indicate how they would rate each experience for the patient on a scale from 0 (terrible experience) to 10 (almost perfect experience). The total score ranges between 0 and 100, with higher scores indicating a better quality of the dying experience.

CONTACTS AND LOCATIONS:
Overall Officials: Sigrun Vehling, PhD, Principal Investigator — Universitätsklinikum Hamburg-Eppendorf
Locations (5):
- Germany (5):
  - Center for Oncology, University Medical Center Hamburg-Eppendorf, Hamburg, Germany
  - Albertinen Krankenhaus, Hamburg, Germany
  - LungenClinic Grosshansdorf, Hamburg, Hamburg
  - Gynecological Outpatient Clinic, University Medical Center Hamburg-Eppendorf, Hamburg
  - Specialized Outpatient Clinic for Autoimmune Liver Disease and for Liver and Bile Duct Tumors, University Medical Center Hamburg-Eppendorf, Hamburg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Philipp R, Kalender A, Harter M, Bokemeyer C, Oechsle K, Koch U, Vehling S. Existential distress in patients with advanced cancer and their caregivers: study protocol of a longitudinal cohort study. BMJ Open. 2021 Apr 24;11(4):e046351. doi: 10.1136/bmjopen-2020-046351. PMID 33895716